CLINICAL TRIAL: NCT05965791
Title: Electrophysiological Assessment of the Median Nerve During the Phalen's Test for Carpal Tunnel Syndrome
Brief Title: Median Nerve Function During Phalen's Test
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: OT-PT-001
Record Dates: First submitted 2023-07-20; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: 30 healthy adult participants aged 18-45 years performing the Phalen's wrist flexion test
  Interventions: Diagnostic Test: Phalen's wrist flexion test

INTERVENTIONS:
Diagnostic Test: Phalen's wrist flexion test — The Phalen's test will be performed at different wrist flexion angles from 0 to 90 degrees.

SUMMARY:
This study will use electromyography and nerve conduction studies to evaluate median nerve function during the Phalen's wrist flexion test in different wrist positions.

DETAILED DESCRIPTION:
The Phalen's test is commonly used to assess carpal tunnel syndrome. However, it is unclear which wrist position during this test best isolates median nerve function. This study will measure thenar muscle activation and median nerve conduction in 30 healthy participants performing the Phalen's test. Different wrist flexion angles will be evaluated to determine which position optimally targets the median nerve. Results may enhance utilization of the Phalen's test in clinical practice and research.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18-45 years
* No history of hand/wrist disorders

Exclusion Criteria:

* Contraindications to EMG or NCV
* Neurological or muscular disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women aged 18-45 recruited from the local community.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-11-25 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Thenar Muscle Activation | Baseline
  Mean EMG activity of the thenar muscles during the Phalen's test at different wrist angles. Measured in microvolts (μV).
Median Nerve Conduction Velocity during Phalen's Test | Baseline
  Median nerve conduction velocity (measured in meters per second, m/s) assessed using surface electrodes at the wrist and elbow during the Phalen's test wrist flexion maneuver. Measured bilaterally at each wrist flexion angle during a single study visit.
Median Nerve Distal Latency during Phalen's Test | Baseline
  Median nerve distal latency (measured in milliseconds, ms) assessed using surface electrodes over the abductor pollicis brevis and stimulating the median nerve at the wrist during the Phalen's test. Measured bilaterally at each wrist flexion angle during a single study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Chair — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No